CLINICAL TRIAL: NCT00001869
Title: Lymphangioleiomyomatosis (LAM) Registry
Brief Title: Official Record of Patients Diagnosed With Lymphangioleiomyomatosis (LAM)
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 990020; 99-H-0020
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2003-04

CONDITIONS: Leiomyomatosis
Keywords: Progesterone; Pulmonary Function Tests; Pneumothorax; Oopherectomy; High Resolution CT; Tuberous Sclerosis Complex; Lymphangioleiomyomatosis (LAM)
MeSH Terms: conditions — Leiomyomatosis; Pneumothorax; Tuberous Sclerosis; Lymphangioleiomyomatosis

SUMMARY:
Pulmonary lymphoangioleiomyomatosis (LAM) is a rare destructive lung disease typically affecting women of childbearing age. Currently, there is no effective therapy for the disease and the prognosis is poor.

In order to better study this disease, the National Heart, Lung, and Blood Institute (NHLBI) has developed a registry to keep an official record of patients diagnosed with LAM. This research project will collect data from 6 health care centers as well as outside physicians. Researchers hope to provide valuable information about the rate of lung destruction and quality of life in patients with LAM.

Patients participating in this study will be followed for 5 years. Tissue collected from these patients may contribute to the development of future studies on the disease processes of LAM.

DETAILED DESCRIPTION:
LAM is a rare disease that predominantly affects women of child-bearing age. To study in more detail this rare disease, this multi-center project will establish a registry of persons with LAM. By combining data from 6 centers and outside physicians, this study may yield valuable information regarding the rate of decline in pulmonary function and quality of life in individuals with LAM. These patients will be followed over a five-year period. Tissue collected from study participants may facilitate future studies into the molecular basis of LAM.

ELIGIBILITY:
Informed consent must be obtained from the patient.

Patients must be female.

Patients must be age 18 or older.

Patients with prevalent and incident cases are eligible.

Patients with the presence or absence of underlying diagnosis or evidence of Tuberous Sclerosis Complex (TSC) are eligible.

Patients must have a diagnosis of LAM confirmed by any of the following criteria:

Lung biopsy (transbronchial, surgical, transthoracic) judged to be diagnostic by the Tissue Core pathologists;

OR

Biopsy of lymph node or other mass judged to be diagnostic by the Tissue Core pathologists;

OR

High resolution CT scan of the chest which is judged to be diagnostic of LAM with a high degree of certainty by all three of the expert radiologists making up the Imaging Core.

Patients may be enrolled in other protocols.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 400
Dates: Start 1998-12; Study Completion 2003-04

CONTACTS AND LOCATIONS:
Locations (1):
- National Heart, Lung and Blood Institute (NHLBI), Bethesda, Maryland, United States

REFERENCES:
- [Background] Abdulla M, Bui HX, del Rosario AD, Wolf BC, Ross JS. Renal angiomyolipoma. DNA content and immunohistochemical study of classic and multicentric variants. Arch Pathol Lab Med. 1994 Jul;118(7):735-9. PMID 8024411
- [Background] Aberle DR, Hansell DM, Brown K, Tashkin DP. Lymphangiomyomatosis: CT, chest radiographic, and functional correlations. Radiology. 1990 Aug;176(2):381-7. doi: 10.1148/radiology.176.2.2367651.
- [Background] Basset F, Soler P, Marsac J, Corrin B. Pulmonary lymphangiomyomatosis: three new cases studied with electron microscopy. Cancer. 1976 Dec;38(6):2357-66. doi: 10.1002/1097-0142(197612)38:63.0.co;2-a. PMID 1000470